CLINICAL TRIAL: NCT01548638
Title: The Effect of the Acetylcholinesterase Inhibitor, Galantamine, on Short-term Abstinence
Brief Title: Effect of Galantamine on Smoking Abstinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 814947
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Nicotine Addiction
Keywords: Tobacco; Smoking; Galantamine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Galantamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Galantamine ER (Experimental): The study will be performed using the 8mg and 16mg doses of galantamine hydrobromide-ER, which is currently marketed for the treatment of Alzheimer's disease.
  Interventions: Drug: Galantamine ER

INTERVENTIONS:
Drug: Galantamine ER — The study will be performed using the 8mg and 16mg doses of galantamine hydrobromide-ER, which is currently marketed for the treatment of Alzheimer's disease. The dosing regimen, which follows FDA-approved guidelines, will be an initial 4 weeks of drug run-up at the lowest 8mg daily dose, followed by an additional one week of drug run-up at the higher dose of 16mg daily.
  Participants will continue to take the 16mg daily during the 7-day quit week, for a total of 6 weeks of treatment with galantamine-ER.
  Other Names: Razadyne ER

SUMMARY:
This is a preliminary open-label study to determine whether a medication called galantamine (Brand Name: Razadyne) will help smokers quit and whether it reduces cognitive problems that smokers experience during a quit attempt.

DETAILED DESCRIPTION:
Galantamine, an FDA-approved treatment for Alzheimer's disease, is used to treat cognitive impairment by enhancing acetylcholine through inhibition of the enzyme, acetylcholinesterase. We propose an open-label pilot feasibility study of short-term (6 weeks) treatment with galantamine.

Sixteen chronic smokers will undergo a validated procedure for screening new medications. Following an initial 4-week drug run-up phase (8mg daily of galantamine-ER), medication dose will be increased to 16 mg daily of galantamine-ER during the fifth and sixth weeks of the study. At the beginning of Week 6, smokers will receive brief counseling and make a 7-day quit attempt.

Following completion of the study, participants will be offered standard smoking cessation treatment. Subjects will perform a working memory task (Visual/Spatial N-Back), a sustained attention task (Continuous Performance Task; CPT), a recall memory task (Word Recognition), a cognitive flexibility task (Wisconsin Card Sort Test), and a response inhibition task (Stop Signal Task). The primary outcome is the ability to remain abstinent during a 7-day quit attempt. Secondary outcomes include change in cognitive performance, adherence, and side effects.

This pilot study will provide information about the role of the cholinergic system during brief abstinence and whether enhancing acetylcholine reduces abstinence-induced cognitive symptoms that promote smoking relapse. Information obtained in this study may further establish cognitive performance measures as endophenotypes for nicotine dependence.

ELIGIBILITY:
Inclusion Criteria:

1. Smokers who are between 18 and 60 years of age who self-report smoking at least 10 cigarettes (menthol and non-menthol) per day for at least the last 6 months.
2. Healthy as determined by the Study Physician, based on a medical evaluation including medical history and physical examination, and psychiatric evaluation.
3. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and Health Insurance Portability and Accountability Act (HIPAA) form.
4. Women of childbearing potential must consent to use a medically accepted method of birth control while participating in the study (e.g., condoms and spermicide, oral contraceptive, Depo-provera injection, contraceptive patch, tubal ligation).

Exclusion Criteria:

1. Smoking Behavior

   * Use of chewing tobacco, snuff, and/or snus.
   * Current enrollment in a smoking cessation program, or use of other smoking cessation medications in the last month or plans to do either in the next 2 months.
   * Provide a carbon monoxide (CO) breath sample reading less than 10ppm at Medical Screening or Baseline visit.
2. Alcohol/Drugs

   * Lifetime history of substance abuse (other than nicotine) and/or currently receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, stimulants, Phencyclidine (PCP), benzodiazepines, or study prohibited medications/recreational drugs) as determined by self-report during the phone screen and/or through the MINI during the Medical Screening.
   * Current alcohol consumption that exceeds 25 standard drinks/week over the past 6 months.
   * Providing a breath alcohol concentration (BrAC) reading of greater than or equal to 0.01 at Medical Screen or Baseline sessions.
   * A positive urine drug screen for cocaine, amphetamines, methamphetamines, benzodiazepines, PCP, methadone, barbiturates, and opiates at the Medical Screening, Baseline visit, and Testing days.
3. Medical

   * Women who are pregnant, planning a pregnancy in the next 3 months, or lactating; all female subjects of child-bearing potential shall undergo a urine pregnancy test prior to enrollment and must agree in writing to use an approved method of contraception. Pregnancy tests will be conducted at the Medical Screening, Baseline visit, and Testing days.
   * Diagnosis of Alzheimer's Disease or dementia.
   * Current treatment of cancer or diagnosed with cancer (except basal cell carcinoma) in the past 6 months.
   * Liver/kidney failure, peptic ulcer disease, benign prostate hypertrophy
   * Asthma or chronic obstructive pulmonary disease (COPD)
   * History (last 6 months) of abnormal heart rhythms, tachycardia and/or cardiovascular disease (stroke, angina, heart attack).
   * Serious or unstable disease within the past 6 months, as determined by the Study Physician.
   * Any impairment (physical and/or neurological) including visual or other impairment preventing cognitive task performance.
   * Uncontrolled high blood pressure (systolic>150 or diastolic>90)
   * Hearing impairment, significant hearing loss (more than 20% in either ear), cochlear implants, or bi-lateral hearing aids.
   * History of brain injury.
   * History of epilepsy or a seizure disorder.
   * Color Blindness.
   * Low or borderline intellectual functioning - determined by receiving a score of less than 90 on the Shipley Institute of Living Scale (SILS) which correlates with the Wechsler Adult Intelligence Scale-Revised (WAIS-R) Estimated Intelligence Quotient (IQ) Test (administered at Medical Screening).
4. Psychiatric Exclusion (as determined by self-report on phone screen and/or through MINI during Medical Screening)

   * Current diagnosis of major depression. Persons with a history of major depression, in remission for 6 months or longer, are eligible, provided they are not excluded based on medications (below).
   * Suicide risk score on MINI greater than 0.
   * History or current diagnosis of schizophrenia, psychosis, or bipolar disorder.
   * Current or past hypomanic/manic episode.
   * Current or history of a diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD).
5. Medication

   * Current use, recent discontinuation (within the last month) of any form of smoking cessation medications (i.e., Zyban, Wellbutrin, Wellbutrin sustained-release (SR), Chantix, nicotine replacement therapy).
   * Current use, recent discontinuation (within the last 60 days) or planned use of the following medications:
   * Anti-anxiety or panic disorder medications.
   * Anti-psychotic medications.
   * Mood-stabilizers (Lithium, Lamictal/lamotrigine, Neurontin/gabapentin, Topamax/topiramate, valproic acid, Tegretol/carbamazepine)
   * Anti-depressants (e.g., Wellbutrin, monoamine oxidase inhibitor (MAOIs), selective serotonin reuptake inhibitor (SSRIs), tricyclic antidepressants).
   * Prescription stimulants (e.g., Provigil, Ritalin, Adderall).
   * Systemic Steroids (e.g., Prednisone).
   * Current use (or use in the past 60 days) of:
   * Alzheimer's disease medications (e.g., Acetylcholinesterase inhibitors (ACIs), Aricept/donepezil, Exelon/rivastigmine, Tacrine, or memantine).
   * Parkinson's disease medications(e.g., Cogentin/benztropine).
   * Irritable bowel syndrome medication (e.g., Dicylomine/Bentyl).
   * Heart medications (e.g., quinidine or Procardia/nifedipine).
   * Peptic ulcer disease medication (e.g, Zantac/ranitidine).
   * Muscle relaxants (e.g., Soma/carisoprodol, Anectine/succinylcholine).
   * Anti-fungal medication (e.g., Nizoral/ketoconazole).
   * Anti-seizure medications (e.g., Ativan, Banzel, Carbatrol, Dilantin, Lamictal, Gabitril, Lyrica, Neurontin, Tegretol, Topamax).
   * COPD medication (e.g., Atrovent/Ipratropium Bromide).
   * Blood pressure medication (e.g., Inversine/Mecamylamine).
   * Urinary retention medications (Duvoid/bethanechol, Proscar/finasteride, Avodart/dutasteride, Dibenzyline/phenoxybenzamine, Regitine/phentolamine).
   * Eye medication (e.g., Atropine).
   * Daily use of:
   * Opiate-containing medications for chronic pain (Duragesic/fentanyl patches, Percocet, Oxycontin).
   * Medication for asthma (albuterol, Serevent, Combivent, Advair, Flovent, Azmacort, Symbicort).
   * Known allergy to study medication.
   * Participants shall be instructed to refrain from using any study prohibited drugs (note - participants are allowed to take prescription medicines not in the exclusion list) throughout their participation in the study.
6. General Exclusion

   * Current enrollment or plans to enroll in another research program in the next 2 months.
   * Any medical condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
   * Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator.
   * Completion of cognitive testing in studies in our center within the last 6 months.
   * Able to effectively communicate in English (reading, writing, speaking).
   * Missing 2 or more consecutive sessions, or 3 or more sessions during the medication period.
   * Missing 2 or more consecutive doses during the medication period.
   * Missing 3 or more doses throughout the medication period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Ashare, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, School of Medicine, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Center for Interdisciplinary Research on Nicotine Addiction homepage — http://www.med.upenn.edu/cirna/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, since recruitment was initiated in March, 2012, 49 (45%) of the 109 completed phone screens resulted in a subject eligible for Intake. Of these subjects, 41 (84%) scheduled an in-person screening visit at our center.
Pre-assignment Details: Of the 29 subjects (73%) who attended the initial eligibility visit, 5 withdrew post enrollment (at visit), 11 were ineligible, and 13 subjects were deemed eligible.
Groups:
- Galantamine ER: The study will be performed using the 8mg and 16mg doses of galantamine hydrobromide-ER, which is currently marketed for the treatment of Alzheimer's disease.
  Galantamine ER : The study will be performed using the 8mg and 16mg doses of galantamine hydrobromide-ER, which is currently marketed for the treatment of Alzheimer's disease. The dosing regimen, which follows FDA-approved guidelines, will be an initial 4 weeks of drug run-up at the lowest 8mg daily dose, followed by an additional one week of drug run-up at the higher dose of 16mg daily.
  Participants will continue to take the 16mg daily during the 7-day quit week, for a total of 6 weeks of treatment with galantamine-ER.
Period: Overall Study
Arm/Group | Galantamine ER
Started | 13
Completed | 9
Not Completed | 4
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Galantamine ER
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Days of Abstinence During a 7-day Quit Attempt
Description: Participants will undergo a 6-week study medication period. Day 36 will be the beginning of a 7-day practice quit attempt, during which number of days of abstinence will be assessed.
Time Frame: Days 36-43; following a 5-week dose run-up
Measure: Mean (Full Range); unit: days
Arm/Group | Galantamine ER
Number analyzed (Participants) | 9
days | 5 [0 to 7]

2. Secondary Outcome: Cognitive Performance: Working Memory Reaction Time
Description: Participants will complete neurocognitive test designed to test working memory and attention and are similar to computer games, in that participants will push a button in response to the pictures they see. Working memory was measured using a computerized N-back task. During the N-back, participants are instructed to remember the location of a stimulus, a grey circle that is approximately 5 cm in diameter, as it appears randomly in 8 possible locations around the perimeter of a computer screen. Stimulus duration is 200 ms, followed by an interstimulus interval (ISI) of 2800 ms. The N-back task includes 4 conditions of varying difficulty levels: the 0-back, 1-back, 2-back, and 3-back.
  Median reaction time to correct responses is described below.
  Typical responses range from 250 ms to 1500 ms.
Time Frame: At Baseline (Day 0), Day 35 (Day before Target Quit Day), and Day 43
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Galantamine ER
Number analyzed (Participants) | 9
ms
  Working Memory Reaction Time Baseline | 575 (122)
  Working Memory Reaction Time Day 35 | 641 (141)
  Working Memory Reaction Time Day 43 | 709 (158)

3. Secondary Outcome: Cognitive Performance: Working Memory Accuracy
Description: Participants will complete neurocognitive test designed to test working memory and attention and are similar to computer games, in that participants will push a button in response to the pictures they see. Working memory was measured using a computerized N-back task. During the N-back, participants are instructed to remember the location of a stimulus, a grey circle that is approximately 5 cm in diameter, as it appears randomly in 8 possible locations around the perimeter of a computer screen. Stimulus duration is 200 ms, followed by an interstimulus interval (ISI) of 2800 ms. The N-back task includes 4 conditions of varying difficulty levels: the 0-back, 1-back, 2-back, and 3-back.
  Number of correct responses (true positives) is described below.
  The maximum number of correct responses is 60.
Time Frame: At Baseline (Day 0), Day 35 (Day before Target Quit Day), and Day 43
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Galantamine ER
Number analyzed (Participants) | 9
correct responses
  Working Memory Accuracy Baseline | 46 (6.6)
  Working Memory Day 35 | 47.4 (7.7)
  Working Memory Day 43 | 46.7 (7.9)

4. Secondary Outcome: Subjective Symptoms (Smoking Urges)
Description: During each visit, we asked subjects to complete the Questionnaire for Smoking Urges-Brief (QSU-B). This measure is an index of urges to smoke, or cigarette craving. The subjective symptoms listed above will be assessed at the following in-person sessions: Baseline session, Days 7, 14, 21, and 28 (brief monitoring visits), Day 35 (Day before Target Quit Day), and Days 37, 39, and 43 (during the 7-day quit attempt).
  The range of possible scores on the QSU-B is 10-70, with higher values indicating increased urges to smoke. This range of scores represents a "total" score; there are no subscales.
Time Frame: Days 7, 14, 21, 28, 35, and 43; Baseline session
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Galantamine ER: The study will be performed using the 8mg and 16mg doses of galantamine hydrobromide-ER, which is currently marketed for the treatment of Alzheimer's disease.
  Galantamine ER: The study will be performed using the 8mg and 16mg doses of galantamine hydrobromide-ER, which is currently marketed for the treatment of Alzheimer's disease. The dosing regimen, which follows FDA-approved guidelines, will be an initial 4 weeks of drug run-up at the lowest 8mg daily dose, followed by an additional one week of drug run-up at the higher dose of 16mg daily.
  Participants will continue to take the 16mg daily during the 7-day quit week, for a total of 6 weeks of treatment with galantamine-ER.
Arm/Group | Galantamine ER
Number analyzed (Participants) | 9
units on a scale
  Baseline | 30.3 (13.9)
  Day 7 | 22.3 (9.4)
  Day 14 | 17 (8.5)
  Day 21 | 20.7 (12.6)
  Day 28 | 21.5 (11.4)
  Day 35 | 34.1 (16.8)
  Day 37 | 21.3 (11.0)
  Day 39 | 19.5 (12.4)
  Day 43 | 17.5 (8.9)

5. Secondary Outcome: Side Effects of Galantamine
Description: Side effects of galantamine were assessed at the following in-person sessions: Baseline session, Days 7, 14, 21, and 28 (brief monitoring visits), Day 35 (Day before Target Quit Day), and Days 37, 39, and 43 (during the 7-day quit attempt). A 37-item checklist of side effects based on the product insert (e.g., Nausea, Vomiting, Diarrhea, Loss of appetite, Stomach pain, Constipation, Gastroesophageal Reflux Problems (Heartburn)) was administered to participants at all study visits after the Intake. An open-ended side effects question was also be included.
  Items were measured on a scale from 0 (None) to 3 (Severe).
  The side effect summary score (total side effects averaged from the 37 item checklist) at each visit is reported below. Each score ranges from 0 (None) to 3 (Severe).
Time Frame: Days 7, 14, 21, 28, 35, 37, 39, and 43; Baseline session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine ER
Number analyzed (Participants) | 9
units on a scale
  Baseline | 0.086 (0.11)
  Day 7 | 0.13 (0.21)
  Day 14 | 0.068 (0.12)
  Day 21 | 0.073 (0.093)
  Day 28 | 0.057 (0.098)
  Day 35 | 0.11 (0.19)
  Day 37 | 0.042 (0.059)
  Day 39 | 0.07 (0.075)
  Day 43 | 0.06 (0.042)

6. Secondary Outcome: Subjective Symptoms (Negative Affect)
Description: Subjects were asked to complete the Positive and Negative Affect Scale (PANAS) to assess symptoms of negative affect (the positive affect scale was not administered). This 10-item scale assesses was assessed at the following in-person sessions: Baseline session, Days 7, 14, 21, and 28 (brief monitoring visits), Day 35 (Day before Target Quit Day), and Days 37, 39, and 43 (during the 7-day quit attempt).
  The range of possible total scores on the PANAS negative affect scale is 10-50, with higher values indicating an increased nicotine withdrawal. This range of scores represent a "total" score; there are no subscales within the negative affect scale of the PANAS.
Time Frame: Days 7, 14, 21, 28, 35, and 43; Baseline session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine ER
Number analyzed (Participants) | 9
units on a scale
  Baseline | 11.4 (1.2)
  Day 7 | 10.1 (.35)
  Day 14 | 10.6 (.74)
  Day 21 | 10.0 (0.48)
  Day 28 | 14.8 (8.3)
  Day 35 | 11.1 (1.5)
  Day 37 | 11.2 (1.6)
  Day 39 | 12.5 (4.4)
  Day 43 | 11.3 (2.1)

7. Secondary Outcome: Subjective Symptoms (Nicotine Withdrawal)
Description: Subjects were asked to complete the Minnesota Nicotine Withdrawal Scale - Revised version (MNWS). The scale assesses eight DSM-IV items of nicotine withdrawal. The subjective symptoms listed above were assessed at the following in-person sessions: Baseline session, Days 7, 14, 21, and 28 (brief monitoring visits), Day 35 (Day before Target Quit Day), and Days 37, 39, and 43 (during the 7-day quit attempt).
  The range of possible total scores on the MNWS is 0-60, with higher values indicating an increased nicotine withdrawal. This range of scores represent a "total" score; there are no subscales.
Time Frame: Days 7, 14, 21, 28, 35, and 43; Baseline session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine ER
Number analyzed (Participants) | 9
units on a scale
  Baseline | 4.3 (1.9)
  Day 7 | 4.3 (2.3)
  Day 14 | 3 (2.4)
  Day 21 | 3.9 (2.8)
  Day 28 | 3.2 (2.6)
  Day 35 | 7 (8.1)
  Day 37 | 4 (3.4)
  Day 39 | 4.9 (4.1)
  Day 43 | 2.4 (2.1)

ADVERSE EVENTS:
Arm/Group | Galantamine ER
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes